CLINICAL TRIAL: NCT01490476
Title: A Single Arm, Single Center, Phase II Trial of RAD001 as Monotherapy in the Treatment of Neurofibromatosis Type 2 - Related Vestibular Schwannoma
Brief Title: Efficacy and Safety Study of RAD001 in the Growth of the Vestibular Schwannoma(s) in Neurofibromatosis 2 (NF2) Patients
Acronym: AFINF2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P101202; 2011-002228-42 (EudraCT Number)
Record Dates: First submitted 2011-11-30; First posted 2011-12-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Neurofibromatosis 2
Keywords: Neurofibromatosis Type 2 with Vestibular Schwannoma; Vestibular Schwannoma; Peripheral Nervous System Diseases; Otorhinolaryngologic Diseases; Vestibulocochlear Nerve Diseases
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic; Peripheral Nervous System Diseases; Otorhinolaryngologic Diseases; Vestibulocochlear Nerve Diseases | interventions — Everolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): Patient with Neurofibromatosis Type 2 and Vestibular Schwannoma treated with RAD001.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — 10 mg per os / day or 05mg per os / day with 12 month
  Other Names: Afinitor / rapamycin

SUMMARY:
The purpose of the study is to determine if RAD001 treatment will shrink or slow the growth of the vestibular schwannoma(s) in Neurofibromatosis 2 (NF2) patients.

DETAILED DESCRIPTION:
This protocol is a Phase II, open-label, efficacy and safety study of single-agent RAD001 in patients with NF2. During the study, subjects will receive continuous daily oral treatment with RAD001 for up to 4 years or until tumor progression.

Primary Objective: To determine whether RAD001 has an effect on the VS growth in patients with NF2 at a rate sufficient to submit the drug for further testing.

Secondary Objectives: To determine whether RAD001 has an effect on the volume of other intracranial tumors; to assess the effect of RAD001 on hearing function in patients with NF2 (when applicable); to determine whether RAD001 modulates signaling pathways in intracranial NF2 tumors removed during the course of the study. And determine the long term safety.

All patients will be treated with RAD001 10 mg p.o. daily dose (5mg if 15-17 years old with cutaneous surface area <1.5m2) for one year except in case of unacceptable toxicity, death, or discontinuation from the study for any other reason.

At 12 months an extension for another one year of RAD001 treatment will be discussed in case of response.

If the patient is stable (decrease or increase lower than 20%), treatment should be stopped and the patient should be kept under quarterly continuous surveillance. Resumption of treatment will be discussed case by case basis if tumor regrowth over 20% relative to the tumor volume at the end of treatment.

All patients will have a follow-up visit (including MRI) scheduled at 24 months after enrollment.

We modify the protocol to extend the treatment by RAD001 for a period of two additional years for stable patients still on treatment two years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NF2 by National Institutes of Health (NIH) criteria
* Age ≥ 15 years
* Progressive VS growth during the previous 12 months. Evidence of disease progression defined by progressive VS during the previous 12 months (>20% increase in volume) in subjects who are at elevated risk for surgical complications (eg, deafness, lower cranial nerve injury, facial weakness) or who refuse surgery
* Adequate bone marrow, liver and renal function.
* For women of childbearing potential, no pregnancy or breast-feeding
* Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Willingness to provide informed consent

Exclusion Criteria:

* Inability to tolerate periodic MRI scans or gadolinium contrast.
* Inability to tolerate periodic audiologic testing or to understand a language with established scoring for word recognition testing.
* Inability to adequately perform volumetric measurement of at least 1 target lesionNote: Patients with cochlear or auditory brainstem implants may participate if a target lesion can be accurately assessed.
* Radiation therapy for the target lesion in the 60 months preceding inclusion in the study.
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug.
* Immunization with attenuated live vaccines within one week of study entry or during study period.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions.
* Patients with a known hypersensitivity to everolimus or other types of rapamycin or to its excipients.
* Patients unwilling to or unable to comply with the protocol

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
effect of RAD001 on the VS growth by MRI | 1 year
  To determine whether RAD001 has an effect on the VS growth in patients with NF2 at a rate sufficient to submit the drug for further testing

SECONDARY OUTCOMES:
Effect of RAD001 on the volume of other intracranial tumors (MRI) and on hearing function (audiogram) | 1, 2 and 4 years after inclusion in the study
  To determine if RAD001 has an effect on the volume of other intracranial tumors, to assess efficacy of RAD001 on hearing function, to determine whether RAD001 modulates signaling pathways in tumors removed during the course of the study and to determine long term safety

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kalamarides, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, 100 boulevard du Général Leclerc, Clichy, France

REFERENCES:
- [Background] Goutagny S, Raymond E, Esposito-Farese M, Trunet S, Mawrin C, Bernardeschi D, Larroque B, Sterkers O, Giovannini M, Kalamarides M. Phase II study of mTORC1 inhibition by everolimus in neurofibromatosis type 2 patients with growing vestibular schwannomas. J Neurooncol. 2015 Apr;122(2):313-20. doi: 10.1007/s11060-014-1710-0. Epub 2015 Jan 8. PMID 25567352